CLINICAL TRIAL: NCT06414473
Title: Sub-Lingual Administration of Cannabidiol for Knee Osteoarthritis
Brief Title: CBD for Knee Osteoarthritis
Acronym: SLACK-OA
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: University of Florida (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: IRB202301136
Record Dates: First submitted 2024-04-24; First posted 2024-05-16 (Actual); Last update posted 2025-09-17 (Actual); Status verified 2025-09

CONDITIONS: Osteoarthritis, Knee
Keywords: Cannabidiol; Osteoarthritis; Pain; Dysfunction; Physical Activity
MeSH Terms: conditions — Osteoarthritis, Knee; Osteoarthritis; Pain; Motor Activity | interventions — Cannabidiol

STUDY DESIGN:
Intervention Model Description: Randomized, double-blind, placebo-controlled, clinical trial
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: All participants, investigators, and study personnel will be blinded to treatment order assignments throughout the study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Active Drug (Active Comparator): Hemp supplement is a full spectrum CBD-rich formulation (~10%) containing very low levels of THC (<0.3%), along with all naturally occurring minor cannabinoids, terpenes, and essential oils from the plant extract.
  Interventions: Drug: Cannabidiol (CBD) Extract
- Vehicle Control (Placebo Comparator): A medium chain triglyceride-based mixing agent blended with coconut oil will be used as the placebo.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Cannabidiol (CBD) Extract — Administered thrice daily (with food) using a sublingual route of administration
  Other Names: Hemp Supplement
  Arms: Active Drug
Drug: Placebo — Administered thrice daily (with food) using a sublingual route of administration
  Other Names: Vehicle Control
  Arms: Vehicle Control

SUMMARY:
Osteoarthritis is a disease that affects millions of Americans and is the leading cause of persistent pain and physical disability in the older adult population. Many physically active Americans have reported pain-relieving effects of cannabidiol (CBD) that can reduce or eliminate use of nonsteroidal anti-inflammatory drugs (NSAIDs) for activity-related pain with minimal to no side effects. Long-term use of over-the-counter medications, including NSAIDs, can pose a significant health risk, and therefore clinical research on the safety and efficacy of CBD is needed.

DETAILED DESCRIPTION:
Knee OA is the most common joint disease and a major cause of functional limitation and pain in adults. Pain is the primary symptom of OA, and the main reason people seek medical treatment. Although pharmacologic treatment for OA such as opioid-based medications may help in the short-term with reducing pain-related symptoms, they are known to have mild to severe side effects along with the potential for long-term dependency. Consequently, many Americans have turned to cannabis-related products like cannabidiol or CBD for reducing pain and pain-related symptoms associated with OA. Current research has shown evidence that phyto-cannabinoids may have a promising therapeutic potential in a variety of physical and psychological ailments, and cannabidiol (CBD) is of particular interest due to its positive safety profile, non-intoxicating effects, and purported therapeutic capabilities in several musculoskeletal diseases. In vitro and in vivo studies have shown that CBD administration in the short term is safe and effective in reducing inflammation and pain behaviors in animal models of OA. Despite the widespread popularity of CBD in the US, there is very limited data that indicates the safety, acceptability, and pain-relieving effects of CBD use for people with symptomatic knee osteoarthritis. The investigators' objective will be to conduct an early-stage clinical trial to investigate the safety, tolerability/acceptability, and efficacy of CBD as a non-pharmacological treatment for symptomatic knee OA. The investigators will conduct an innovative and novel study with rigorous scientific design that will assess and monitor symptomatic relief and improved function following CBD administration (active) or placebo-control using a randomized, double-blind, placebo-controlled, cross-over study design. The investigators will be recruiting 30 adult men and women, between 40 and 75 years of age, with an established clinical diagnosis of knee OA. To be included in the study, participants must report having moderate to severe knee pain (≥4/10) with physical activity in one or both knees. Subjects will be required to complete a 78-day study trial spanning a pre-dosing screening visit, baseline testing, 30-day dosing regimen with follow-up testing. A 2-week wash-out period will be followed by the cross-over phase using identical baseline and follow-up testing procedures. The data from the active CBD phase will be compared to data from the placebo-control phase. There is an extremely large consumer base for CBD-related products in the US, and this base will be expanding exponentially over the course of this decade; therefore, scientific investigation into its therapeutic potential is necessary.

ELIGIBILITY:
Inclusion Criteria:

1. established clinical diagnosis of knee osteoarthritis (KOA)
2. moderate to severe knee pain (≥4/10) with physical activity in one or both knees

Exclusion Criteria:

1. pregnant (urine pregnancy test) or lactating
2. current cannabis (THC and/or CBD) use (urine drug screen)
3. any prior or ongoing medical condition that, in the investigators' opinion, could adversely affect the safety of the subject
4. any major surgery within 3 months prior to recruitment or planned orthopedic surgery for any time during this study which would interfere with the ability to report pain or quality of life outcome measures
5. any exposure to another investigational drug within 3 months prior to screening
6. BMI ≥ 45
7. current use of any enzyme-modifying drugs, including strong inhibitors or strong inducers of cytochrome P (CYP) enzymes
8. history of:

   1. suicidal ideation or self-harm behavior
   2. seizure disorder or traumatic brain injury,
   3. liver or kidney disease, and
   4. cardiovascular diseases

Ages: 40 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2024-06-14 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Patient-Reported Outcomes version of the Common Terminology Criteria for Adverse Events (PRO-CTCAE) | Weekly until 1 month
  Categorical scale, None or not at all (0) and very severe or very much (4), higher scores mean worse outcome
Theoretical Framework of Acceptability Questionnaire (TFAQ) | Baseline and 1 month
  Likert scale, 1 and 5, higher scores mean worse outcome
Self-report Ratings of Knee Pain | Baseline and 1 month, daily until 1 month
  Numeric Rating Scale, 0 and 10, higher scores mean worse outcome
Physical Activity | Daily until 1 month
  Accelerometer measures step counts per day
Western Ontario and McMaster Universities Arthritis Index (WOMAC) | Baseline and 1 month
  Categorical scale, none (0) and extreme (4), higher scores mean worse outcome

SECONDARY OUTCOMES:
Quantitative Sensory Testing (QST) | Baseline and 1 month
  A set of noninvasive tests used to assess pain sensitivity
Physical Function | Baseline and 1 month
  Timed Stair-climbing Test (sec)
Fear of Pain Questionnaire III (FPQ III) | Baseline and 1 month
  Likert scale, 0 and 5, higher scores mean worse outcome
Pain Catastrophizing Scale (PCS) | Baseline and 1 month
  Likert scale, 0 and 4, higher scores mean worse outcome
Pain Anxiety Symptom Scale (PASS-20) | Baseline and 1 month
  Likert scale, 0 and 5, higher scores mean worse outcome
Pittsburgh Sleep Quality Index (PSQI) | Baseline and 1 month
  Categorical scale, Not during the past month to and Three or more times a week, higher scores mean worse outcome

CONTACTS AND LOCATIONS:
Locations (1):
- Sports Medicine Research Laboratory, Gainesville, Florida, United States